CLINICAL TRIAL: NCT06962514
Title: Effects of Low Load Resistance Exercise With a Blood Flow Restriction Cuff on Strength, Balance, Physical Performance, Depression and Cognition in Older Adults: a Randomized Controlled Double-blind Study
Brief Title: Low Load With Blood Flow Restriction for Improving Strength, Balance, and Cognition in Older Adults
Acronym: BFRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Hongje Jang, Physical Therapist, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-07-005-009
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Blood Flow Restriction Exercise; Resistance Training; Elderly (People Aged 65 or More); Muscle Strength; Balance; Cognition; Depression
Keywords: Blood flow restriction training; Older adults; Muscle mass; Functional Mobility; Cognition
MeSH Terms: conditions — Depression | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two-group parallel randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors were blinded to group assignment. Both groups followed the same exercise protocol, and the use of BFR cuffs was not disclosed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BFR group (Experimental): Exercise with BFR cuff
  Interventions: Other: Blood flow restriction cuff
- Exercise group (Experimental): Exercise without BFR cuff
  Interventions: Other: Exercise without BFR cuff

INTERVENTIONS:
Other: Blood flow restriction cuff — Use of blood flow restriction cuff during resistance training. The cuff pressure is set at 50% of the participant's arterial occlusion pressure.
  Arms: BFR group
Other: Exercise without BFR cuff — Resistance exercise performed without blood flow restriction. Same protocol as BFR group but without cuff application.
  Arms: Exercise group

SUMMARY:
This study aims to examine the effects of low load resistance exercise with a blood flow restriction cuff on muscle strength, balance, physical performance, depression, and cognitive function in community-dwelling older adults.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the effects of low-load resistance exercise combined with blood flow restriction (BFR) in community-dwelling older adults. A total of 26 participants aged 65 and older will be randomly assigned to either a BFR exercise group or a control group that performs the same resistance exercises without BFR.

The intervention will be conducted twice a week for 8 weeks (16 sessions total). The BFR cuffs will be applied at 50% of the participant's arterial occlusion pressure. Both groups will undergo the same exercise protocol, supervised by trained personnel. Assessments will be performed at baseline and after the intervention.

Primary outcome measures include lower limb strength (5 Times Sit-to-Stand Test), balance ability (Timed Up and Go test), gait performance (10-meter walk test, GaitRite), muscle mass index (SMI) using BWA 2.0, muscle thickness (quadriceps via ultrasound), cognitive function (MoCA), depression level (GDS-K).

Both participants and outcome assessors are blinded to group allocation. This study has received IRB approval from Sahmyook University Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling individuals aged 65 years and older who have not had a fall in the past year.
2. No neurological or musculoskeletal condition that would interfere with exercise performance.
3. Clear consciousness and able to communicate effectively.
4. Capable of reading and writing.
5. Able to understand the research explanation and provide informed consent.

Exclusion Criteria:

1. Orthopedic, neurological, or vascular conditions that may affect vital signs such as dizziness, blood pressure instability, or fall risk during assessment.
2. Any history of musculoskeletal surgery within the past 6 months.
3. Physician-determined health status that contraindicates exercise participation.
4. Cognitive or literacy impairments that hinder understanding of study procedures.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Quadriceps muscle thickness (via ultrasound) | From baseline to the end of the 8-week intervention.
  Muscle thickness of the rectus femoris and vastus intermedius will be assessed using B-mode ultrasound at rest. Measurements will be taken pre- and post-intervention.
Skeletal Muscle Mass Index (SMI) | From baseline to the end of the 8-week intervention.
  SMI will be calculated using appendicular lean mass obtained from bioelectrical impedance analysis (BWA 2.0) and height squared (kg/m²). Handgrip strength will also be assessed as an indicator of muscle function.

SECONDARY OUTCOMES:
Lower limb strength (5 Times Sit to Stand Test) | From baseline to the end of the 8-week intervention.
  Lower extremity strength will be assessed using the Five Times Sit to Stand Test, measuring the time required to stand from a chair and sit down five times.
Depression level (GDS-K) | From baseline to the end of the 8-week intervention.
  Depressive symptoms will be assessed using the Korean version of the Geriatric Depression Scale (GDS-K), a standardized self-report screening tool for older adults. It consists of 30 items, each answered with "Yes" or "No." The total score ranges from 0 to 30, with higher scores indicating more severe depressive symptoms. Scores are interpreted as follows: 0-13 = normal, 14-18 = mild depression, 19-21 = moderate depression, and 22 or above = severe depression.
Cognitive function (MoCA) | From baseline to the end of the 8-week intervention.
  Cognitive function will be evaluated using the Korean version of the Montreal Cognitive Assessment (MoCA-K), a validated screening tool for mild cognitive impairment in older adults. It assesses multiple cognitive domains, including attention, memory, language, visuospatial skills, executive functions, and orientation. The total score ranges from 0 to 30, with higher scores indicating better cognitive performance. A score below 23 is generally considered indicative of cognitive impairment. One point may be added for individuals with 6 or fewer years of formal education.
Gait performance (10-meter walk test and Gaitrite) | From baseline to the end of the 8-week intervention.
  Gait speed and spatiotemporal gait parameters will be measured using a 10-meter walk test and GaitRite system at comfortable walking speed.
Balance ability (TUG) | From baseline to the end of the 8-week intervention.
  Dynamic balance will be assessed using the Timed Up and Go (TUG) test.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahmyook University, Graduate School of Physical Therapy, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) has not been finalized. The data may be considered for sharing after de-identification and upon request, depending on future publication requirements and institutional policy.